CLINICAL TRIAL: NCT02584244
Title: Feasibility of the LUM Imaging System for Detection of Gastrointestinal Cancers
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lumicell, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LUM-015/2.6-002; P50CA127003 (NIH)
Record Dates: First submitted 2015-10-16; First posted 2015-10-22 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Cancer; Pancreatic Cancer; Esophageal Cancer; Gastric Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms; Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Six groups enrolling up to 11 patients each. Groups are patients with colorectal cancer, patients with esophageal cancer, patients with pancreatic cancer receiving neoadjuvant chemotherapy, patients with pancreatic cancer not receiving neoadjuvant chemotherapy, gastric cancer patients who have received neoadjuvant therapy, and patients with early stage gastric cancer or precancerous lesions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (6):
- Patients with colorectal cancer (Experimental): The first 3 patients will be injected at a dose of 0.5 mg/kg. If no or minimal activity is observed and no serious adverse events occur, the subsequent three patients will be injected with the second tier dose level of 1.0 mg/kg. If no or minimal activity is observed in in the second tier dosing group, and no serious adverse events occur, the following three patients will have the third tier dose of 1.5 mg/kg administered. An additional 2 patients will be recruited at the dose level that produces optimal LUM015 activity. All surgical specimens will be sent to the pathology suite for imaging with the LUM 2.6 Imaging Device and routine diagnostic assessment.
  Interventions: Drug: LUM015; Device: LUM 2.6 Imaging Device
- Patients with esophageal cancer (Experimental): The first 3 patients will be injected at a dose of 0.5 mg/kg. If no or minimal activity is observed and no serious adverse events occur, the subsequent three patients will be injected with the second tier dose level of 1.0 mg/kg. If no or minimal activity is observed in in the second tier dosing group, and no serious adverse events occur, the following three patients will have the third tier dose of 1.5 mg/kg administered. An additional 2 patients will be recruited at the dose level that produces optimal LUM015 activity. All surgical specimens will be sent to the pathology suite for imaging with the LUM 2.6 Imaging Device and routine diagnostic assessment.
  Interventions: Drug: LUM015; Device: LUM 2.6 Imaging Device
- Pancreatic cancer patients receiving neoadjuvant chemotherapy (Experimental): The first 3 patients will be injected at a dose of 0.5 mg/kg. If no or minimal activity is observed and no serious adverse events occur, the subsequent three patients will be injected with the second tier dose level of 1.0 mg/kg. If no or minimal activity is observed in in the second tier dosing group, and no serious adverse events occur, the following three patients will have the third tier dose of 1.5 mg/kg administered. An additional 2 patients will be recruited at the dose level that produces optimal LUM015 activity. All surgical specimens will be sent to the pathology suite for imaging with the LUM 2.6 Imaging Device and routine diagnostic assessment.
  Interventions: Drug: LUM015; Device: LUM 2.6 Imaging Device
- Pancreatic cancer patients not receiving neoadjuvant chemo (Experimental): The first 3 patients will be injected at a dose of 0.5 mg/kg. If no or minimal activity is observed and no serious adverse events occur, the subsequent three patients will be injected with the second tier dose level of 1.0 mg/kg. If no or minimal activity is observed in in the second tier dosing group, and no serious adverse events occur, the following three patients will have the third tier dose of 1.5 mg/kg administered. An additional 2 patients will be recruited at the dose level that produces optimal LUM015 activity. All surgical specimens will be sent to the pathology suite for imaging with the LUM 2.6 Imaging Device and routine diagnostic assessment.
  Interventions: Drug: LUM015; Device: LUM 2.6 Imaging Device
- Gastric cancer patients who have received neoadjuvant therapy (Experimental): The first 3 patients will be injected at a dose of 0.5 mg/kg. If no or minimal activity is observed and no serious adverse events occur, the subsequent three patients will be injected with the second tier dose level of 1.0 mg/kg. If no or minimal activity is observed in in the second tier dosing group, and no serious adverse events occur, the following three patients will have the third tier dose of 1.5 mg/kg administered. An additional 2 patients will be recruited at the dose level that produces optimal LUM015 activity. All surgical specimens will be sent to the pathology suite for imaging with the LUM 2.6 Imaging Device and routine diagnostic assessment.
  Interventions: Drug: LUM015; Device: LUM 2.6 Imaging Device
- Patients with early stage gastric cancer or precancerous lesions (Experimental): The first 3 patients will be injected at a dose of 0.5 mg/kg. If no or minimal activity is observed and no serious adverse events occur, the subsequent three patients will be injected with the second tier dose level of 1.0 mg/kg. If no or minimal activity is observed in in the second tier dosing group, and no serious adverse events occur, the following three patients will have the third tier dose of 1.5 mg/kg administered. An additional 2 patients will be recruited at the dose level that produces optimal LUM015 activity. All surgical specimens will be sent to the pathology suite for imaging with the LUM 2.6 Imaging Device and routine diagnostic assessment.
  Interventions: Drug: LUM015; Device: LUM 2.6 Imaging Device

INTERVENTIONS:
Drug: LUM015
Device: LUM 2.6 Imaging Device

SUMMARY:
The overall goal of this feasibility study is to assess the initial safety and efficacy of LUM015 in ex vivo far-red imaging of colorectal, pancreatic, and esophageal cancers (adenocarcinoma) using the LUM Imaging System.

DETAILED DESCRIPTION:
The overall goal of this feasibility study is to assess the initial safety and efficacy of a novel, intravenously administered cathepsin activatable imaging probe, LUM015, in ex vivo far-red imaging of colorectal, pancreatic, and esophageal cancers (adenocarcinoma) using the LUM Imaging Device.

All subjects will have an established diagnosis of colorectal, pancreatic, or esophageal adenocarcinoma and are scheduled for resection of their primary tumors.

Patients will be seen by their surgeon or endoscopist in an office visit and undergo routine preoperative testing within eight weeks of their planned procedure. During the pre-procedure visit a complete history and physical examination and standard of care pre-operative laboratory studies (including ECG) will be performed. These laboratory values and results of the history and physical will be used to confirm eligibility. For some patients, a pre-procedure visit is not required as part of standard treatment. Those patients may have a study-specific screening and pre-procedure laboratory tests at their local medical center. On the day of their planned surgery, LUM015 will be administered by bolus intravenous injection. For colorectal and esophageal cases, LUM015 will be administered 2-6 hours prior to tumor resection. For pancreatic cases, given the variability in predicting the time to tumor resection relative to surgical start time, injection will occur 1 hour prior to planned surgical start time. Patients will be monitored for adverse events until discharged from the hospital. Follow up of subjects will continue until their first post-operative visit.

All surgical specimens (whether containing normal tissue or tumor tissue) will be sent to the pathology suite for imaging with the LUM Imaging Device and routine diagnostic assessment. Imaged areas showing high fluorescence will be marked to guide pathology evaluation and determine whether the area contains tumor. Samples of imaged areas showing low fluorescence signal will also be evaluated by pathology to determine whether the area only contains normal tissue. After imaging, part of this tissue will be fresh frozen for correlative studies.

The patients are expected to be admitted to the hospital for the surgical procedure and remain in the hospital post-surgery as indicated and required by the surgeon per standard of care treatment. While in the hospital, patients will be assessed for adverse events. Laboratory studies will also be performed during this time as a part of routine post-surgical care and to assess for any imaging agent related adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histologically or cytologically confirmed esophageal, colorectal or pancreatic adenocarcinoma (inclusive of high grade dysplasia and cystic neoplasms) on a biopsy prior to surgery and must be scheduled for surgical resection, inclusive of endoscopic mucosal resection, of the primary tumor. Subjects at any cancer stage will be enrolled.
2. Subjects may have previously received pre-operative radiation therapy and neoadjuvant chemotherapy.
3. Age of 18 years or older.
4. Subjects must be able and willing to follow study procedures and instructions.
5. Subjects must have received and signed an informed consent form.
6. Subjects must be sufficiently healthy to undergo surgery or an endoscopic procedure.
7. Subjects must have normal organ and marrow function as defined below:

   * Leukocytes >/= 3,000/mcL
   * Absolute neutrophil count >/= 1,500/mcL
   * Platelets >/= 100,000/mcL
   * total bilirubin within normal institutional limits (except in cases of malignant biliary obstruction)
   * AST (SGOT)/ALT (SGPT) </= 2.5 X institutional upper limit of normal (</= 5 x ULN in cases of malignant biliary obstruction)
   * Creatinine within normal institutional limits or creatinine clearance >/= 60 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal.
8. Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) starting the day entering the study, and for 60 days after injection of the imaging agent. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
9. Subjects with ECOG performance status of 0 or 1.

Exclusion Criteria:

1. Subjects who have taken an investigational drug within 30 days of enrollment.
2. Subjects with QTc interval > 480ms.
3. Subjects who have not recovered from adverse events due to pharmaceutical or diagnostic agents administered more than 4 weeks earlier.
4. Subjects with uncontrolled hypertension defined as persistent systolic blood pressure > 180 mm Hg, or diastolic blood pressure > 110 mm Hg; those subjects with known HTN should be under these values while under pharmaceutical therapy
5. History of allergic reaction attributed to drugs containing polyethylene glycol (PEG)
6. History of allergic reaction to oral or intravenous contrast agents.
7. Pregnant women or lactating women
8. Subjects who are sexually active and not willing/able to use medically acceptable forms of contraception upon entering the study.
9. HIV-positive individuals on combination antiretroviral therapy.
10. Any subject for whom the investigator feels participation is not in the best interest of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2016-08-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Correlate LUM015 fluorescence in gastrointestinal cancers (pancreatic, esophageal, and colorectal) with pathology results | 1 day

SECONDARY OUTCOMES:
Number of safety events in humans with colorectal, pancreatic, and esophageal cancer. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T Chan, M.D., Ph.D, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States